CLINICAL TRIAL: NCT01599351
Title: Different Radiation Exposures to Patient and Endoscopists Between Performing ERCP in Patients Lying Prone and Left Lateral Decubitus
Brief Title: Radiation Exposure During Endoscopic Retrograde Cholangiopancreatography Between Prone and Left Lateral Decubitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PA-E-RAD001
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Exposure to Ionizing Radiation
Keywords: Radiation exposure; ERCP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prone (Active Comparator): Patients were in prone position along the ERCP procedure.
  Interventions: Radiation: The radiographic-fluoroscopic system
- Left lateral decubitus (Active Comparator): Patients were in left lateral decubitus along the ERCP procedure.
  Interventions: Radiation: The radiographic-fluoroscopic system

INTERVENTIONS:
Radiation: The radiographic-fluoroscopic system — Fluoroscopy was used during ERCP procedure. With automatic brightness adjustment, patients with thicker body will get greater radiation dose.
  Other Names: Siemens Model Polystar

SUMMARY:
The objective of this study is to evaluate the radiation dose to patient at two positions (prone and left lateral) and to medical staff during Endoscopic retrograde cholangiopancreatography (ERCP) procedure using dose area product (DAP) meter and thermoluminescent dosimeter (TLD). Data were recorded on 20 patients at prone position and 20 patients at left lateral position.

DETAILED DESCRIPTION:
The radiographic-fluoroscopic system manufactured by Siemens Model POLYSTAR was used for ERCP procedure at King Chulalongkorn Memorial Hospital. Dose Area Product (DAP) manufactured by PTW Model DIAMENTOR E, a transmission ionization chamber was attached to X-ray collimator to record the dose-area (cGy.cm2) in order to determine the entrance surface air kerma (ESAK, mGy) of the patients at two positions (prone and left lateral) while the Kodak Portal Pack for localization imaging was placed on the patient's couch to determine the exposed area (cm2) on the surface of the patient. TLD was attached at five positions, left eye, thyroid, left forearm, lower abdomen and left leg of the medical staff during ERCP procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with common bile duct (CBD) stone and underwent ERCP
* age over 18 years
* ASA class I-II

Exclusion Criteria:

* Pregnant
* Abnormal coagulation
* ASA class III-IV
* Emergency/urgency conditions
* Unstable vital signs
* Denied to participate the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Patients' entrance surface dose | within 12 hours after procedure
  Transparent ionization chamber was placed at the light beam diaphragm of the x-ray tube to measure the dose in the air and the verification film was placed on the couch at fluoroscopic area to determine exposed area. Patient's dose-area product will express in cGy.cm2.

SECONDARY OUTCOMES:
Endoscopists' radiation dose | Within 12 hours after procedure
  Thermoluminescent dosimeters (TLD) were placed at left eye, thyroid, left forearm, lower abdomen, and left leg of endoscopists. The TLDs used in this study was TLD-100 which was lithium fluoride crystal doped with magnesium and titanium (LiF:Mg, Ti). After procedures all labeled TLDs were read by automatic TLD reader (Harshaw 5500, Thermo Scientific Corp., MA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Phonthep Angsuwatcharakon, MD, MSc, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Patumwan, Bangkok, Thailand